CLINICAL TRIAL: NCT02572349
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IW-1701 Administered Orally as Single Doses to Healthy Subjects
Brief Title: Trial of IW-1701 (A Stimulator of Soluble Guanylate Cyclase (sGC)) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-1701-101
Record Dates: First submitted 2015-10-07; First posted 2015-10-08 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IW-1701 (Experimental): Single Dose
  Interventions: Drug: IW-1701
- Matching Placebo for IW-1701 (Placebo Comparator): Single Dose
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: IW-1701
  Arms: IW-1701
Drug: Matching Placebo
  Arms: Matching Placebo for IW-1701

SUMMARY:
The objectives of the study are to assess the safety and tolerability of a range of single doses of IW-1701 when administered as oral capsules to healthy subjects, to determine the pharmacokinetic profile and pharmacodynamics effects of a range of single doses of IW-1701 when administered as oral capsules to healthy subjects.

ELIGIBILITY:
Inclusion:

* Between 18 and 60 years old at the Screening Visit;
* Women of childbearing potential must have a negative pregnancy test and must agree to use double-barrier contraception;
* BMI > 18.5 and < 32.0 kg/m2 at the Screening Visit;
* In overall good health with no clinically significant laboratory, ECG, or physical exam findings;
* Other inclusion criteria per protocol.

Exclusion:

* History of any clinically-significant medical condition;
* Other exclusion criteria per protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Assessment of the safety and tolerability of IW-1701 in healthy subjects via adverse events | From baseline up to 8 days
  The primary objectives of this study are to assess the safety and tolerability of single ascending dosage levels of IW-1701 versus placebo in healthy subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Ironwood Investigational Site, San Antonio, Texas, United States